CLINICAL TRIAL: NCT05272852
Title: PersAFOne III: Feasibility Study of the FARAPULSE Pulsed Field Ablation System Plus - PersAF in the Treatment of Persistent Atrial Fibrillation
Brief Title: The FARAPULSE PersAFOne III Trial for the Treatment of Persistent Atrial Fibrillation
Acronym: CS1543
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1543
Record Dates: First submitted 2021-12-13; First posted 2022-03-10 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE™ Pulsed Field Ablation System Plus (Experimental): Ablation using FARAPULSE™ Pulsed Field Ablation System Plus
  Interventions: Device: FARAPULSE™ Pulsed Field Ablation System Plus

INTERVENTIONS:
Device: FARAPULSE™ Pulsed Field Ablation System Plus — Ablation using FARAPULSE™ Pulsed Field Ablation System Plus

SUMMARY:
The objective of this safety and feasibility study is to assess whether the endocardial creation of electrically nonconductive lesions via PEF catheter ablation applied using the FARAPULSE Pulsed Field Ablation System Plus-PersAF is a feasible and safe treatment for PersAF and associated AFL

DETAILED DESCRIPTION:
PersAFOne III study is a prospective, multi-center safety and feasibility study in subjects with persistent AF. Subjects will undergo percutaneous PEF ablation for pulmonary vein isolation as well as cavotricuspid isthmus interruption and other left atrial ablations at the investigator's discretion. Subjects will then be followed at 30 days, 60 ± 15 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90 day blanking period and other relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Study subjects are required to meet all the following inclusion criteria to participate in this study:

1. Patients with documented drug-resistant symptomatic persistent AF meeting all three of the following criteria:

   1. Patient is refractory or intolerant to at least one Class I/III antiarrhythmic agent.
   2. ECG-documented first episode of persistent AF, lasting longer than 7 days but not longer than 365 days
   3. Holter within 90 days prior to the Enrollment Date demonstrating 24 hours of continuous AF
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient participation requirements:

   1. Lives locally
   2. Is willing and capable of providing Informed Consent to undergo study procedures
   3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study

      -

Exclusion Criteria:

Subjects will be excluded from participating in this study if they meet any one of the following exclusion criteria:

1. AF that is:

   1. Paroxysmal (longest AF episode < 7days)
   2. Longstanding (has persisted > 12 months or that does not respond to cardioversion if < 12 months)
   3. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
2. Left atrial anteroposterior diameter ≥ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. Hemodynamically significant valvular disease
   3. Prosthetic heart valve
   4. NYHA Class III or IV CHF
   5. Previous endocardial or epicardial ablation or surgery for AF
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial appendage device or occlusion
   9. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
   10. Significant or symptomatic hypotension
   11. Bradycardia or chronotropic incompetence
   12. History of pericarditis
   13. History of rheumatic fever
   14. History of congenital heart disease with any residual anatomic or conduction abnormality
4. Any of the following within 3 months prior toenrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery (e.g. coronary artery bypass grafting, ventriculotomy, atriotomy)
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
5. History of blood clotting or bleeding abnormalities.
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Contraindications to CT or MRI
8. Sensitivity to contrast media not controlled by premedication
9. Women of childbearing potential who are pregnant, lactating or not using birth control
10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to

    1. Body mass index (BMI) > 40
    2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    4. Renal insufficiency with an estimated creatinine clearance <30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
    5. Active malignancy or history of treated cancer within 24 months of enrollment
    6. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    7. Clinically significant infection
    8. Predicted life expectancy less than one year
11. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
12. Current or anticipated enrollment in any other clinical study
13. Employment by FARAPULSE or the same hospital department or office of any investigator, or a family member of any of the preceding groups.
14. Use of amiodarone after day of index ablation procedure. Patients will cease use of amiodarone on or before the date of the index ablation procedure.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, Principal Investigator — Nemocnice Na Homolce (homolka)
Locations (2):
- Czechia (2):
  - Neuron Medical, Brno
  - Nemocnice Na Homolce, Prague

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Started | 80
Completed | 77
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 80

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Composite Safety Endpoint (CSE) Defined as the Incidence of the Following Early-onset and Late-onset Serious Adverse Events (SAEs) Which Are Device- or Procedure-related, as Adjudicated by the CEDMC
Description: Percentage of Intent to Treat subjects with one or more of the specified device or procedure related SAEs Endpoint(CSE) defined as the incidence of the following early-onset serious adverse events (SAEs) which are device- or procedure-related, as adjudicated by the Clinical Events and Data Monitoring Committee (CEDMC). Atrioesophageal fistula and PV stenosis components will be assessed for occurrence at any time during follow-up.
  Early onset (within 30 days of an Index or Remap Procedure)
  * Death
  * Myocardial infarction (MI)
  * Persistent diaphragmatic paralysis
  * Stroke or transient ischemic attack (TIA)
  * Peripheral or organ thromboembolism
  * Pericarditis
  * Cardiac tamponade / perforation
  * Vascular access complications requiring intervention
  * Heart block Late onset (any time during follow-up through 12 months)
  * Pulmonary vein (PV) stenosis (> 70% diameter reduction from baseline)
  * Atrio-esophageal fistula
Time Frame: 30Days-12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants | 1

2. Primary Outcome: Primary Effectiveness Endpoint: Acute Procedural Success Acute Vein Success
Description: Demonstration of Acute Vein Success in all attempted PVs using the FARAPULSE Cardiac Ablation System Plus during the first ablation procedure (Index or Rescheduled Index Procedure)
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 77
Participants | 77

3. Secondary Outcome: The Primary Safety Endpoint Assessed at 7 Days
Description: Percentage of Intent to Treat subjects with one or more of the specified device or procedure related SAEs Endpoint(CSE) defined as the incidence of the following early-onset serious adverse events (SAEs) which are device- or procedure-related, as adjudicated by the Clinical Events and Data Monitoring Committee (CEDMC). Atrioesophageal fistula and PV stenosis components will be assessed for occurrence at any time during follow-up.
  Early onset (within 7 days of an Index or Remap Procedure)
  * Death
  * Myocardial infarction (MI)
  * Persistent diaphragmatic paralysis
  * Stroke or transient ischemic attack (TIA)
  * Peripheral or organ thromboembolism
  * Pericarditis
  * Cardiac tamponade / perforation
  * Vascular access complications requiring intervention
  * Heart block Late onset (any time during follow-up through 12 months)
  * Pulmonary vein (PV) stenosis (> 70% diameter reduction from baseline)
  * Atrio-esophageal fistula
Time Frame: 7-Days
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants | 1

4. Secondary Outcome: The Percentage of Subjects With a Device- or Procedure-related SAE
Description: Percentage of subjects with one or more device or procedure related SAEs.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants
  Device Related Serious Adverse Events (SAEs) | 0
  Procedure Related Serious Adverse Events (SAEs) | 3

5. Secondary Outcome: The Percentage of Subjects With Stroke or TIA
Description: The percentage of occurrence of stroke or TIA observed in any subjects
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants | 0

6. Secondary Outcome: The Percentage of Subjects Requiring Cardioversions
Description: The percentage of subjects where cardioversion (s) was performed within the 12-month post index
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants | 5

7. Secondary Outcome: The Percentage of Subjects Requiring an Arrhythmia-related (AF, AFL or AT) Hospitalization
Description: The percentage of subjects that were hospitalized for arrhythmia-related (AF, AFL or AT) reasons
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
Number analyzed (Participants) | 80
Participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE™ Pulsed Field Ablation System Plus
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 14/80
Other Adverse Events (participants affected / at risk) | 38/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE™ Pulsed Field Ablation System Plus (N=80)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 2 (2)
Blood Pressure Fluctuation (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE™ Pulsed Field Ablation System Plus (N=80)
Arteriospasm coronary (Cardiac disorders) | 15 (15)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 10 (10)
Haemorrhage (Vascular disorders) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT05272852/Prot_SAP_001.pdf